CLINICAL TRIAL: NCT07071844
Title: BEvacizumab Plus Trifluridine/Tipiracil in a Bi-WEEkly Administration to Reduce Grade 3-4 Neutropenia in Patients With mCRC: A Prospective, Multicenter, Comparative, Randomized GERCOR G-124 BETWEEN Phase II Study
Brief Title: BETWEEN: Biweekly Bevacizumab + Trifluridine/Tipiracil to Reduce Grade 3-4 Neutropenia in mCRC Patients
Acronym: BETWEEN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BETWEEN
Record Dates: First submitted 2025-06-19; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Trifluridine/Tipiracil; metastatic colorectal cancer; neutropenia; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Neutropenia | interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is prospective, multicenter, comparative randomized phase II study design to assess the impact of a biweekly administration (experimental Arm A) compared to a conventional administration (control Arm B) on the rate of grade 3-4 neutropenia in metastatic colorectal cancer (mCRC) patients treated with trifluridine/tipiracil plus bevacizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (experimental) - Trifluridine/tipiracil plus bevacizumab biweekly administration (Experimental): Trifluridine/tipiracil: 35 mg/m², twice daily (BId) orally, on days 1-5 and days 15-19; 1 cycle every 28 days.
  + Bevacizumab: 5 mg/kg intravenously (IV) on day 1 and day 15; 1 cycle every 28 days.
  Interventions: Drug: Trifluridine/tipiracil; Drug: Bevacizumab
- Arm B (control) - Trifluridine/tipiracil plus bevacizumab conventional administration (Active Comparator): Trifluridine/tipiracil: 35 mg/m² Bid orally on days 1-5 and days 8-12; 1 cycle every 28 days.
  + Bevacizumab: 5 mg/kg IV on day 1 and day 15; 1 cycle every 28 days.
  Interventions: Drug: Trifluridine/tipiracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Trifluridine/tipiracil — 35 mg/m², orally
  Other Names: LONSURF
Drug: Bevacizumab — 5 mg/kg, intravenous route
  Other Names: AVASTIN

SUMMARY:
This study was design to:

* To assess the impact of a biweekly (experimental arm) compared to a conventional administration (control arm) on the rate of grade 3-4 neutropenia in metastatic colorectal cancer (mCRC) patients treated with trifluridine/tipiracil plus bevacizumab, and
* To identify predictive clinical and biological factors for grade 3-4 neutropenia in this patient population.

DETAILED DESCRIPTION:
Trifluridine/tipiracil is effective in refractory metastatic colorectal cancer (mCRC), as shown in phase III trials, including SUNLIGHT, which demonstrated improved PFS and OS when combined with bevacizumab, setting a new third-line standard. However, this combination raises grade 3-4 neutropenia rates to 43-66%, often leading to dose reductions or delays. A biweekly regimen tested in a small phase II trial showed reduced neutropenia (15.9%) but limited generalizability. Neutropenia remains a major concern, with 9.5% mortality. G-CSF may help manage risk, especially in high-risk patients (LONGBOARD).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent,
2. Patients willing and able to comply with protocol requirements,
3. Age ≥ 18 years,
4. ECOG PS 0-1,
5. Histologically proven colorectal adenocarcinoma,
6. Stage IV disease,
7. Previous chemotherapy regimens with each of the following agents: fluoropyrimidine, oxaliplatin, irinotecan, anti-VEGF therapy (bevacizumab, aflibercept, and anti-EGFR therapy (cetuximab or panitumumab for tumors with RAS and/or BRAF wild-type),
8. Tumor assessment (CT-scan or MRI) no later than 21 days prior to treatment - at least one measurable or evaluable lesion as assessed by computed tomography (CT)-scan or magnetic resonance imaging (MRI) according to RECIST,
9. Known BRAF and RAS mutational status, and microsatellite instability/mismatch repair deficiency (MSI/dMMR) status,
10. Have life expectancy of at least 3 months,
11. Adequate hematologic function: neutrophils >1.5 x 10^9/L; platelets >100 x 10^9/L; hemoglobin ≥ 9 g/dL,
12. Adequate renal function: Calculated (regardless of the calculation method) creatinine clearance (CrCl) ≥30 mL/min), proteinuria < 2+ (dipstick urinalysis) or ≤1g / 24h,
13. Adequate liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit normal (ULN; ≤5 x ULN in case of liver metastasis), total bilirubin ≤1.5 x ULN (<2 x ULN if hyperbilirubinemia is due to Gilbert's syndrome), albumin ≥25 g/L,
14. Clinical and blood baseline evaluations no later than 14 days prior to treatment,
15. Ability to swallow oral tablets,
16. Women must be surgically sterile or postmenopausal, or not be pregnant, breastfeeding, or expecting to conceive during the study. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to starting trifluridine/tipiracil treatment. WOCBP must agree to use an adequate method of contraception or birth control for the duration of study treatment and least 6 months (trifluridine/tipiracil, bevacizumab) after the last dose of the study treatment,
17. Males who are fertile and sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment and at least 6 months (trifluridine/tipiracil, bevacizumab) after the last dose of the study treatment.
18. Is willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study,
19. Registration with the French National Health Care System or PUMA (Protection Universelle Maladie).

Exclusion Criteria:

1. ECOG PS 2,
2. Medical history or evidence of CNS metastasis upon physical examination, unless adequately treated (e.g., non-irradiated CNS metastasis, seizure not controlled with standard medical therapy, patients are stable without evidence of progression for at least 28 days prior to inclusion),
3. Local or locally advanced disease (stage I to III),
4. Concomitant unplanned antitumor therapy (e.g., chemotherapy, molecular targeted therapy, immunotherapy),
5. Unresolved grade ≥3 non-hematologic toxicity related to previous chemotherapy regimen (excluding alopecia and skin pigmentation),
6. Dihydropyrimidine dehydrogenase (DPD) deficiency (uracilemia dosage >16 ng/ml); Uracilemia dosing results must be available before inclusion,
7. Treatment with warfarin,
8. Treatment with any other investigational medicinal product (IMP) within 28 days prior to inclusion,
9. Symptomatic carcinomatosis with occlusive symptoms or ascites requiring paracentesis,
10. Other serious and uncontrolled non-malignant disease (e.g., active infection requiring systemic therapy, coronary stenting or myocardial infarction, or stroke in the past 6 months prior inclusion),
11. Severe or uncontrolled active acute or chronic infection,
12. Major surgery within 28 days (4 weeks) prior to inclusion,
13. Gastrointestinal disease that could potentially interfere with study drug absorption,
14. Uncontrolled diabetes mellitus, hypertension, or cardiac arrhythmia,
15. Active (or history of) interstitial lung disease or pulmonary hypertension,
16. Major adverse cardiovascular event within 6 months prior to inclusion,
17. Severe/unstable angina, or NYHA class III or IV heart failure,
18. Systemic immunosuppressive therapy, except steroids given prophylactically or at chronic low dosage (≤20 mg/day prednisone equivalent),
19. Radiotherapy within 28 days (4 weeks) before randomization, except for palliation,
20. Serious nonhealing wound, ulcer or bone fracture,
21. Deep vein thromboembolic event within 28 days (4 weeks) prior to inclusion,
22. Known clinically relevant coagulopathy, bleeding diathesis or bleeding event within 28 days (4 weeks) prior to inclusion,
23. Malignant disease other than mCRC,
24. Other concomitant or previous malignancy, except i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
25. Rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.

    Note: In patients who have previously received or are receiving intravenous bisphosphonates, invasive dental procedures should be avoided, if possible.

    Note: Caution is required when using medicinal products that are human thymidine kinase substrates, e.g., zidovudine. Such medicinal products, if used concomitantly with trifluridine/tipiracil, may compete with the effector, trifluridine, for activation via thymidine kinases. Therefore, when using antiviral medicinal products that are human thymidine kinase substrates, monitor for possible decreased efficacy of the antiviral medicinal product, and consider switching to an alternative antiviral medicinal product that is not a human thymidine kinase substrate, such as lamivudine, didanosine, and abacavir.

    Note: It is unknown whether trifluridine/tipiracil may reduce the effectiveness of hormonal contraceptives. Therefore, women using hormonal contraceptive must also use a barrier contraceptive method.
26. Human immunodeficiency virus (HIV)-infected patients or otherwise known to be HIV-positive,
27. Untreated hepatitis B virus (HBV) or hepatitis C virus (HCV),
28. Concomitant administration of prophylactic phenytoin and live attenuated virus vaccine such as yellow fever vaccine 28 days (4 weeks) prior to treatment,
29. Impossibility of submitting to the medical follow-up of the study for geographical, social, or psychiatric illness,
30. Under legal protection regime (guardianship, curatorship, judicial safeguard) or administrative decision or incapability of giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The occurrence of at least one grade 3-4 neutropenia | From randomization up to 14 days after the end of treatment
  The occurrence of 3-4 neutropenia in mCRC patients undergoing treatment with the combination of bevacizumab and bi-weekly administration of trifluridine/tipiracil (experimental arm) compared to a conventional administration (control arm).

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death from any cause, assessed up to 3 years
  OS in both arms; calculated from the date of randomization to the date of death from any cause.
Progression-free survival (PFS) | From randomization to the date of the first documented disease progression or death due to any cause, up to 3 years
  PFS in both arms; defined as the time from randomization to the date of the first documented PD determined by the Investigator assessment by RECIST 1.1 or death due to any cause, whichever occurs first
Best overall response (BOR) | From randomization to the date of progression, death or subsequent anti-cancer therapy, up to 3 years
  BOR according to Response Evaluation Criteria Solid Tumors (RECIST) v1.1 in both arms; defined as the best response designation (CR, PR, SD or PD), evaluated on all radiological evaluations available and related to study treatment period.
Disease control rate (DCR) | Up to achievement of best overall response (BOR) of CR or PR or SD, up to 3 years
  DCR in both arms according to RECIST v1.1; defined as at least a CR, PR or SD radiological evaluation designation on all radiological evaluations available and related to study treatment period.
Incidence and grade of adverse events (AEs) and serious adverse events (SAEs) [Safety and tolerability] | Assessed 28 days after the last administration of treatment or after the end of the treatment visit
  Incidence and grade of AEs and SAEs, according to NCI-CTCAE v 5.0 in both arms
Eastern Cooperative Oncology Group performance status (ECOG PS) deterioration | Time from baseline up to 3 years
  ECOG PS deterioration is defined as the first increase of at least one point from baseline. The ECOG PS scale ranges from 0 (fully active, asymptomatic) to 4 (completely bedridden), with higher scores indicating worse functional status and poorer prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste BACHET, MD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (10):
- France (10):
  - CHU Amiens, Amiens
  - Centre Hospitalier Universitaire -Besançon, Besançon
  - Centre François Baclesse, Caen
  - Centre Hospitalier Departemental Vendee - Site Des Oudairies, La Roche-sur-Yon
  - Centre Hospitaler Universitaire de Lille, Lille
  - Hôpital privé Jean MERMOZ, Lyon
  - CHU Saint-Antoine, Paris
  - Institut Saint Catherine, Paris
  - CHU de BORDEAUX Hôpital HAUT-LEVEQUE, Pessac
  - Institut de cancérologie Strasbourg Europe, Strasbourg

IPD SHARING:
Plan to Share IPD: No